CLINICAL TRIAL: NCT04998370
Title: Hemoglobin in the Cerebrospinal Fluid to Monitor for Secondary Brain Injury After Aneurysmal Subarachnoid Hemorrhage - a Prospective Multinational Validation Study
Brief Title: Cerebrospinal Fluid Hemoglobin to Monitor for Aneurysmal Subarachnoid Hemorrhage Related Secondary Brain Injury
Acronym: HeMoVal
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Michael Hugelshofer, Principal Investigator, University of Zurich
Other Study IDs: 2021-01023
Record Dates: First submitted 2021-07-19; First posted 2021-08-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Vasospasm; Delayed Cerebral Ischemia; Delayed Ischemic Neurological Deficit
Keywords: Cerebrospinal Fluid; Hemoglobins
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid supernatant (after centrifugation)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: The study population consists of patients admitted to an academic tertiary care center due to an aneurysmal subarachnoid hemorrhage. The primary objective of the study focuses on patients included with external ventricular drain (EVD), while secondary objectives consider patients with both EVD and lumbar drain (LD) as well as patients without any drainage system.

SUMMARY:
The primary objective of this study is to evaluate the association between hemoglobin levels in the cerebrospinal fluid (CSF-Hb) and the occurrence of secondary brain injury in patients after aneurysmal subarachnoid hemorrhage (SAH-SBI) during the first 14 days after bleeding.

DETAILED DESCRIPTION:
This is an international multicentre observational study to validate cerebrospinal fluid hemoglobin (CSF-Hb) as a monitoring biomarker for aneurysmal subarachnoid hemorrhage related secondary brain injury (SAH-SBI). It is hypothesized that there is an association between the concentration of CSF-Hb and the occurrence of SAH-SBI during the first 14 days after the bleeding (post-SAH).

The primary objective of this study is to evaluate the association between ventricular CSF-Hb and SAH-SBI during the first 14 days post-SAH.

The secondary objectives are to investigate:

* the association between ventricular CSF-Hb and angiographic vasospasms (aVSP), delayed cerebral ischemia (DCI) and delayed ischemic neurological deficits (DIND) during the first 14 days post-SAH,
* the accuracy of ventricular CSF-Hb to monitor for aVSP, DCI and DIND during the first 14 days post-SAH,
* the association between lumbar CSF-Hb and SAH-SBI, aVSP, DCI and DIND during the first 14 days post-SAH,
* the accuracy of lumbar CSF-Hb to monitor for aVSP, DCI and DIND during the first 14 days post-SAH,
* the association between baseline measures and CSF-Hb (ventricular and lumbar during the first 14 days post-SAH),
* the association between CSF-Hb (ventricular and lumbar during the first 14 days post-SAH) and co-interventions/complications,
* the association between CSF-Hb (ventricular and lumbar during the first 14 days post-SAH) and chronic hydrocephalus at 12 weeks follow-up,
* the association between CSF-Hb (ventricular and lumbar during the first 14 days post-SAH) and functional outcome at 12 weeks follow-up,
* exploratory CSF proteome/metabolome analyses to assess Hb toxicity, inflammation, neuronal, or vascular damage.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* hospital admission due to an aneurysmal subarachnoid hemorrhage (diagnosis radiologically confirmed)

Exclusion Criteria:

* non-aneurysmal subarachnoid hemorrhage (eg. trauma, perimesencephalic subarachnoid hemorrhage).
* participation in another study with CSF sampling or an interventional medical product within the 30 days preceding and during the present study.
* previous enrolment into the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients admitted to an academic tertiary care center due to an aneurysmal subarachnoid hemorrhage. The primary objective of the study focuses on patients included with EVD, while secondary objectives consider patients with both, EVD and LD as well as patients without any drainage system.
Sampling Method: Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Aneurysmal subarachnoid hemorrhage related secondary brain injury (SAH-SBI) | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  Composite outcome consisting of angiographic vasospasms (aVSP), delayed cerebral ischemia (DCI), or delayed ischemic neurological deficits (DIND).

SECONDARY OUTCOMES:
Angiographic vasospasms (aVSP) | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  The definition of aVSP comprises a narrowing of cerebral arteries based on a digital subtraction angiography (DSA), CT angiography (CTA) or magnetic resonance angiography (MRA). In the absence of an appropriate imaging procedure on the respective day, this will be noted as no imaging performed.
Delayed cerebral ischemia (DCI) | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  DCI is defined as new ischemia or new infarction on CT/perfusion CT or MRI. In the absence of an appropriate imaging procedure on the respective day, this will be noted as no imaging performed.
Delayed ischemic neurologic deficits (DIND) | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  DIND is defined as a new focal neurological deficit or a decrease in Glasgow Coma Scale (GCS) of at least 2 points for at least 2 hours. In case the patient cannot be clinically assessed (e.g., sedation), this will be noted as non-assessable).
Co-intervention 1: Nimodipine treatment | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  Whether the patient received preventive nimodipine treatment within the past 24 hours.
Co-intervention 2: Spasmolysis | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  Whether a rescue therapy with pharmacological spasmolysis or balloon angioplasty was performed within the past 24 hours.
Co-intervention 3: Intraventricular administration of rtPA (ICV-rtPA) | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  Whether rtPA was administered via the EVD to induce blood clot lysis within the past 24 hours.
Co-intervention 4: Triple-H-therapy | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  A triple-H-therapy or elements of it (hypertension, hypervolemia or hemodilution) was induced within the past 24 hours.
Co-intervention 5: Decompression | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  A surgical decompression (e.g. decompressive hemicraniectomy) was performed within the past 24 hours.
Complication 1: CSF infection | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  Differentiated between infection (Clinical symptoms and signs of CSF infection and positive CSF culture), colonization (2 positive CSF cultures without clinical symptoms and signs) and contamination (1 positive CSF culture with consecutive culture being negative).
Complication 2: Surgical site infection | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  Evidence for a surgical site infection at the EVD/LD skin entrance site.
Chronic hydrocephalus | 12 weeks follow-up visit
Functional status 1: Glasgow Outcome Scale Extended [1-8] | 12 weeks follow-up visit
  1. Death
  2. Vegetative state (unresponsive and speechless)
  3. Lower severe disability (requires frequent help of someone to be around at home most of the time every day)
  4. Upper severe diasbility (can be left alone > 8h during the day, but unable to travel and/or go shopping without assistance)
  5. Lower moderate disability (unable to work or only in sheltered workshop)
  6. Upper moderate disability (reduced work capacity; resumes <50% of the pre-injury level of social and leisure activities)
  7. Lower good recovery (minor problems that affect daily life; resumes >50% of the pre-injury level of social and leisure activities)
  8. Upper good recovery (no current problems related to the brain injury that affect daily life)
Functional status 2: modified Rankin Scale [0-6] | 12 weeks follow-up visit
  0 No symptoms
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some helpt, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead

OTHER OUTCOMES:
Cerebrospinal fluid hemoglobin | Day 1 to day 14 after the aneurysmal subarachnoid hemorrhage
  CSF sampling: CSF sampling will be performed via EVD or LD, depending on the patient's access to the CSF space. The decision regarding the insertion of an EVD or LD is made independently of this study and according to the clinical standard of care. 2ml of CSF will be sampled on a daily basis at approximately the same time in the morning.
  CSF centrifugation and storage: Immediately after sample collection, the CSF will be centrifuged at 1500 G for 15 minutes. The cell-free CSF supernatant will be stored at -80°C until analysis.
  Spectrophotometric cerebrospinal fluid hemoglobin (CSF-Hb) measurements: Absorption spectra in the visual range between 350 and 650 nm of all CSF samples will be measured. Quantification of oxyhemoglobin in CSF (CSF-Hb) will be performed using spectral deconvolution.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hugelshofer, MD MSc, Principal Investigator — University Hospital and University of Zurich, Department of Neurosurgery; Kevin Akeret, MD/PhD, Principal Investigator — University Hospital and University of Zurich, Department of Neurosurgery; Dominik J Schaer, MD, Study Chair — University Hospital and University of Zurich, Department of Internal Medicine; Raphael M Buzzi, MD/PhD, Study Chair — University Hospital and University of Zurich, Department of Internal Medicine
Locations (8):
- Austria (2):
  - Johannes Kepler Universität Linz, Universitätsklinik für Neurochirurgie, Linz
  - Medizinische Universität Wien, Klinik für Neurochirurgie, Vienna
- Germany (3):
  - Universitätsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Klinikum rechts der Isar TUM, München, Bavaria
  - Universitätsklinikum Tübingen, Tübingen, Tübingen
- Switzerland (3):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - University Hospital Zurich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Akeret K, Buzzi RM, Saxenhofer M, Bieri K, Chiavi D, Thomson BR, Gruttner-Durmaz M, Schwendinger N, Humar R, Regli L, van Doormaal TPC, Held U, Keller E, Hugelshofer M, Schaer DJ; HeMoVal Research Group. The HeMoVal study protocol: a prospective international multicenter cohort study to validate cerebrospinal fluid hemoglobin as a monitoring biomarker for aneurysmal subarachnoid hemorrhage related secondary brain injury. BMC Neurol. 2022 Jul 18;22(1):267. doi: 10.1186/s12883-022-02789-w. PMID 35850705